CLINICAL TRIAL: NCT04516135
Title: A Randomized Phase II Trial of Palliative Pelvic Radiation Therapy to Improve Health Related Quality of Life in Gynecologic Malignancies
Brief Title: Single Fraction or Multi-fraction Palliative Radiation Therapy for the Improvement of Quality of Life in Patients With Metastatic Gynecologic Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0517; NCI-2020-05684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0517 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (radiation therapy) (Experimental): Patients undergo standard of care radiation therapy in the form of 3D CRT, IMRT, or VMAT at the physician's discretion for 1 fraction in the absence of disease progression or unacceptable toxicity. Patients with < 30% decrease in the SIS may receive an additional fraction on day 21 at the physician's discretion.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Volume Modulated Arc Therapy
- Arm B (radiation therapy) (Active Comparator): Patients undergo standard of care radiation therapy in the form of 3D CRT, IMRT, or VMAT at the physician's discretion over 2 weeks for 10 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Volume Modulated Arc Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D CRT
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Volume Modulated Arc Therapy — Undergo VMAT
  Other Names: VMAT

SUMMARY:
This phase II trial studies if a single session of palliative radiation therapy can help improve symptoms of gynecologic cancers that have spread to other places in the body (metastatic) and that affect quality of life as well or more so than multiple sessions (which is the standard of care). Palliative radiation therapy may help patients with metastatic gynecologic cancers live more comfortably. Researchers also want to learn how radiation affects the immune system and to compare the effects of giving one radiation treatment to giving multiple radiation treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether single fraction palliative radiation therapy (SFRT) improves health-related quality of life (HR-QOL) over multi-fraction palliative radiotherapy (MFRT).

SECONDARY OBJECTIVES:

I. To determine whether single fraction palliative radiation therapy (SFRT) improves individual domains of health-related quality of life (HR-QOL) over multi-fraction palliative radiotherapy (MFRT).

II. To determine whether SFRT increases clinically meaningful HR-QOL improvement over MFRT.

III. To determine whether SFRT provides non-inferior symptom burden improvement to MFRT.

IV. To describe radiation related toxicity rates within 21 days and within year for patients receiving SFRT and MFRT.

EXPLORATORY OBJECTIVES:

I. To describe T-cell repertoire of patients receiving SFRT and MFRT. II. To describe vaginal microbiome of patients receiving SFRT and MFRT. III. To describe gut microbiome of patients receiving SFRT and MFRT. IV. To describe financial burden of patients undergoing palliative pelvic radiation with either SFRT or MFRT.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo standard of care radiation therapy in the form of 3-dimensional conformal radiation therapy (3D CRT), intensity-modulated radiation therapy (IMRT), or volume modulated arc therapy (VMAT) at the physician's discretion for 1 fraction in the absence of disease progression or unacceptable toxicity. Patients with < 30% decrease in the Symptom Inventory Scale (SIS) may receive an additional fraction on day 21 at the physician's discretion.

ARM B: Patients undergo standard of care radiation therapy in the form of 3D CRT, IMRT, or VMAT at the physician's discretion over 2 weeks for 10 fractions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented gynecologic cancer with prior or current evidence of metastatic disease
* Measurable pelvic disease with any pain and/or bleeding
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3
* Estimated life expectancy > 3 months at discretion of treating physician
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication
* Patient able to provide properly obtained written informed consent
* Gynecologic Section Radiation Oncology Quality Assurance (QA) for eligibility for single fraction radiation treatment

Exclusion Criteria:

* Prior pelvic radiation therapy that would make treatment unsafe at the discretion of the treating physician
* Systemic therapy concurrently or within 21 days of first dose of radiation
* Concurrent participation in another interventional radiation therapy trial concurrently or within 30 days of study consent. Note: Patients who are participating in systemic clinical trials and non-interventional clinical trials (e.g., QOL, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation
* Known second malignancy that requires active treatment (at the discretion of the primary investigator)
* Documented psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding at any point starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change in index value of EuroQol 5 Dimensions - 5 Levels (EQ-5D-5L) score | Baseline up to 21 days post-radiation therapy
  An index value will be calculated for each participant according to page 13 of the user guide. Scores will be summarized using descriptive statistics. Will use a 2-sample t-test to compare the change scores between the single fraction palliative radiation therapy (SFRT) and multi-fraction palliative radiation therapy (MFRT) groups.

SECONDARY OUTCOMES:
Absolute change in mobility | Baseline up to 21 days post-radiation therapy
  Each dimension is rated on a scale from 1 to 5 where 1 represents no problem present or patient can care for self and 5 represents extreme problems present or unable to care for self. Improvement within each dimension will be assessed by the absolute change of heath state. A decrease in the raw score by 1 or more points denotes improvement within the dimension.
Absolute change in self-care | Baseline up to 21 days post-radiation therapy
  Each dimension is rated on a scale from 1 to 5 where 1 represents no problem present or patient can care for self and 5 represents extreme problems present or unable to care for self. Improvement within each dimension will be assessed by the absolute change of heath state. A decrease in the raw score by 1 or more points denotes improvement within the dimension.
Absolute change in activity | Baseline up to 21 days post-radiation therapy
  Each dimension is rated on a scale from 1 to 5 where 1 represents no problem present or patient can care for self and 5 represents extreme problems present or unable to care for self. Improvement within each dimension will be assessed by the absolute change of heath state. A decrease in the raw score by 1 or more points denotes improvement within the dimension.
Absolute change in pain | Baseline up to 21 days post-radiation therapy
  Each dimension is rated on a scale from 1 to 5 where 1 represents no problem present or patient can care for self and 5 represents extreme problems present or unable to care for self. Improvement within each dimension will be assessed by the absolute change of heath state. A decrease in the raw score by 1 or more points denotes improvement within the dimension.
Absolute change in anxiety | Baseline up to 21 days post-radiation therapy
  Each dimension is rated on a scale from 1 to 5 where 1 represents no problem present or patient can care for self and 5 represents extreme problems present or unable to care for self. Improvement within each dimension will be assessed by the absolute change of heath state. A decrease in the raw score by 1 or more points denotes improvement within the dimension.
>= 6 point increase in EuroQol-Visual Analogue Scale | Baseline up to 21 days post-radiation therapy
  Will summarize the number of patients with clinical meaningful health-related (HR)-quality of life (QOL) improvement using frequencies and proportions. The proportion of patients with clinically meaningful HR-QOL improvement will be compared between SFRT and MFRT using a chi-squared test.
Decrease in Symptom Inventory (SIS) | At 21 days post-radiation therapy
  Will be calculated as the average of the worst pain, least pain, pain on average, pain right now and scores from the vaginal bleeding questions. The change in SIS score from baseline to 21 days post radiation therapy will be calculated for each patient and evaluated between the SFRT and MFRT groups using a t-test. Will be calculated as the average of the worst pain, least pain, pain on average, pain right now and scores from the vaginal bleeding questions. The change in SIS score from baseline to 21 days post radiation therapy will be calculated for each patient and evaluated between the SFRT and MFRT groups using a t-test.
Incidence of adverse events | Within 21 days and up to 1 year
  Assessed per Common Terminology Criteria for Adverse Events version 5.0. Radiation related toxicity event rates within 21 days and within one year for patients receiving SFRT and MFRT will be summarized using frequencies and proportions. Proportions between SFRT and MFRT will be compared using a chi-squared or Fisher's exact test.

OTHER OUTCOMES:
T-cell repertoire | Up to 1 year
  Will describe T-cell clonality, diversity, clonal overlap, productive and nonproductive frequencies using descriptive statistics. Informal comparisons may be completed to generate hypotheses for future studies.
Vaginal microbiome | Up to 1 year
  Will use alpha and beta diversity metrics for both 16S and whole-genome sequencing (WGS), including overall diversity, richness and evenness and species-specific microbial dynamics. Will be summarized using descriptive statistics. Informal comparisons may be completed to generate hypotheses for future studies.
Gut microbiome | Up to 1 year
  Will use alpha and beta diversity metrics for both 16S and WGS sequencing, including overall diversity, richness and evenness and species-specific microbial dynamics. Will be summarized using descriptive statistics. Informal comparisons may be completed to generate hypotheses for future studies.
Financial burden | Up to 21 days
  Will be assessed using the Economic Strain and Resilience in Cancer Financial Toxicity Questionnaire. The scores for each question will be summarized using descriptive statistics. An overall average score will be calculated by calculating the mean score of the seven questions. At the end of the questionnaire, the patient is asked to rate their overall financial situation as much better, better, nearly the same, worse, or much worse. The frequency of each answer to the global question will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Colbert, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Cooper Hospital University, Camden, New Jersey
  - OhioHealth, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org